CLINICAL TRIAL: NCT01267032
Title: Improving Smoking Cessation Outcomes in PTSD With CBT for Insomnia
Brief Title: Helping Veterans Quit Smoking by Improving Their Sleep
Acronym: ISCWCBTI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated after two years by CSRD
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPLA-09-S09; 1I01CX000301-01 (Other Grant/Funding Number: DVA)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Delivery of Health Care, Integrated; Desensitization, Immunologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Integrated Care + Cognitive-Behavioral Treatment for Insomnia
  Interventions: Behavioral: Integrated Care; Behavioral: Cognitive-Behavioral Treatment for Insomnia
- Arm 2 (Sham Comparator): Integrated Care + Desensitization Treatment for Insomnia
  Interventions: Behavioral: Integrated Care; Behavioral: Desensitization Treatment for Insomnia

INTERVENTIONS:
Behavioral: Integrated Care — A PTSD-aware smoking cessation intervention developed by Miles McFall, PhD.
Behavioral: Cognitive-Behavioral Treatment for Insomnia — A behavioral treatment aimed at improving sleep continuity and subjective sleep through stimulus control, sleep restriction, and attenuation of maladaptive sleep-related cognitions.
  Arms: Arm 1
Behavioral: Desensitization Treatment for Insomnia — A credible sham treatment for insomnia matching CBTI in treatment time, patient expectations, therapist expectations, etc.
  Arms: Arm 2

SUMMARY:
This project is designed to determine whether an efficacious behavioral intervention for insomnia can improve the quit rates achieved by an efficacious smoking cessation program aimed at PTSD patients ("Integrated Care"). A second aim is to deepen our understanding of the mechanisms relating sleep and smoking in PTSD.

DETAILED DESCRIPTION:
In summary, participation will involve a screening period of approximately one week, six weeks of temporally aligned IC ("Integrated Care" - manualized smoking cessation treatment integrating components of behavioral treatment for PTSD) and behavioral sleep treatments (Cognitive-Behavioral Treatment for Insomnia or CBTI), and follow-up telephone interviews at two months and six months.

Screening: Patients in the VA Palo Alto inpatient psychiatry and domiciliary programs indicating interest in quitting cigarette smoking will be pre-screened by the Medical Director to determine whether an individual's psychiatric conditions contraindicates use of bupropion or NRT (Nicoderm). Patients interested in quitting will be referred to the study coordinator. Coordinator will be notified whether medication or NRT is contraindicated for participant and/or of a diagnosed sleep disorder (treated or untreated) other than insomnia.

Continuing participants will be consented and then complete 24 hours of cued symptom reporting using a personal digital assistant (PDA) to verify their capacity to adhere to this component of the study protocol. Continuing participants will undergo a research psychodiagnostic assessment followed by an ambulatory screening polysomnogram (PSG) to exclude undiagnosed sleep disorders. (Participants exhibiting evidence of sleep disorder will be referred for a clinical sleep study.) Screening assessments and psychodiagnostics have been sequenced with the aim of minimizing burden for those excluded.

Participants meeting all inclusion and exclusion criteria will be randomized to IC+CBTI or IC+Desensitization Treatment for Insomnia (DTI: a manualized placebo control intervention). They will meet twice with the IC therapist to complete IC sessions 1 and 2. Over the course of these sessions, they will negotiate a quit date at least three weeks from that time and at least four weeks prior to their projected discharge from inpatient treatment. (Inpatient stays in both of these programs average thirteen weeks.) IC sessions 3 and 4 will be evenly spaced between IC session 2 and the planned quit date. Three weeks prior to their quit date, they will initiate sleep treatment (sessions 1 and 2) and nightly mattress actigraphy. Two weeks prior to their quit date they will begin PDA-based EMA. One to two weeks prior to their quit date, they will commence bupropion and receive sleep treatment session 3. One week prior to their quit date they will receive sleep treatment session 4. On their quit date they will begin NRT. Thereafter, for weeks four through six, they will receive IC sessions five through eight and sleep treatment session five through seven, respectively. At the end of week six, they will receive IC session eight which will also serve as the 3 week assessment of smoking status (the primary outcome assessment of the study). (Note that the first planned assessment of cessation status will occur prior to the expected discharge date for all participants.) The final research interventions will be telephone interviews at two months and six months. Salivary cotinine samples will be obtained at the end of each post-quit week (only if the participant is not using NRT) the last corresponding to the primary outcome assessment, at both telephone follow-up smoking status assessments (by mail).

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be smokers who have smoked at least 10 cigarettes per day for the past year,
* are motivated to make a smoking cessation attempt,
* are na ve to behavioral sleep treatment and are willing to be randomly assigned to either one of the sleep treatment arms.
* Participants must meet the criteria for PTSD and or partial PTSD.
* They will indicate a willingness to forgo the use of all alternative tobacco products during their attempt to quit cigarettes.
* They will be fluent in English.

Exclusion Criteria:

* Candidates who meet DSM-IV criteria for schizophrenia,
* current manic syndrome,
* lifetime but not current PTSD or partial PTSD,
* or current substance abuse/dependence will be excluded.
* positive Brain Injury Screen will not result in exclusion from the study.
* subjects reporting a prior diagnosis of severe obstructive sleep apnea will be excluded unless they have been successfully treated via weight loss, surgery, or continuous positive airway pressure to which they are reliably adherent.
* We expect these criteria to exclude 15 to 20% of potential participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
seven-day point prevalence abstinence | 21 days post-quit-day

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Woodward, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States